CLINICAL TRIAL: NCT06194578
Title: A Phase 0, Single-Center Study to Evaluate the Safety and Tolerability of Injecting Sterile Saline Subcutaneously Into the Abdomen and Thigh of Healthy Volunteers Using Varying Volumes and Rates of Infusion
Brief Title: A Study of Sterile Saline Infusion in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-TEC-275823
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subcutaneous Infusion of Sterile Saline (Experimental): Participants will receive sterile saline subcutaneous infusion administered into abdomen and/or anterior thigh through various sizes of needles at various volume and rate of delivery at Visit 1.
  Interventions: Other: Sterile Saline

INTERVENTIONS:
Other: Sterile Saline — Sterile saline will be administered subcutaneously.

SUMMARY:
The purpose of the study is to evaluate the influence of needle size, injected fluid volume, and rate of fluid on the degree of pain experienced by adult healthy volunteers after subcutaneous infusion of sterile saline.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than (>)18 and less than (<) 36
* Able to understand the English language
* Has a negative coronavirus-2019 (COVID-19) test result at the time of admission, prior to administration of study intervention

Exclusion Criteria:

* Age < 18 years and > 60 years
* BMI < 18 or > 36
* Unable to understand the English language
* Currently pregnant or lactating
* History of skin sensitivity or allergy to steel needle or adhesive tape
* History of abnormal blood coagulation or bleeding
* History of abnormal immune function or frequent skin infections
* Active cardiovascular, pulmonary, dermatologic, endocrine, rheumatologic, hematologic, ophthalmologic, psychiatric, metabolic, hepatic, renal, immune, gastrointestinal, neurological, or musculoskeletal disease
* Has tattoo(s) or scarring at the site of injection or any other condition which may interfere with the injection site examination, in the opinion of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Participant's Pain Intensity as Assessed by Visual Analog Scale (VAS) Score | Up to 10 minutes after completion of the saline infusion
  Participant's pain intensity during or after the saline infusion as assessed by VAS score will be reported. VAS is a self-reported pain rating scale ranging 0=no pain to 100=worst possible pain.
Participant's Pain Intensity as Assessed by Verbal Pain Score (VPS) | Up to 10 minutes after completion of the saline solution
  Participant's pain intensity during or after the saline infusion as assessed by VPS will be reported. VPS will be graded by participants as none, mild, moderate, and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency